CLINICAL TRIAL: NCT01315093
Title: Role of Heparin in Poor Responders Undergoing In Vitro Fertilisation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Assistant Professor, Director of the ARU, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2011-03-08; First posted 2011-03-15 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2016-03

CONDITIONS: Infertility
Keywords: In Vitro Fertilisation; poor responders
MeSH Terms: conditions — Infertility | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Heparin, Low-Molecular-Weight group (Experimental): LMWH was administered during an IVF cycle using either the GnRH - agonist or antagonist protocol in poor responders. Drug was started at the beginning of the cycle and stopped at the time of pregnancy test if negative, or continued if pregnancy occurred until the 32th weeks of gestation
  Interventions: Drug: Heparin, Low-Molecular-Weight
- Non Heparin, Low-Molecular-Weight group (Active Comparator): IVF cycle using either the GnRH - agonist or antagonist protocol in poor responders.
  Interventions: Drug: no heparin

INTERVENTIONS:
Drug: Heparin, Low-Molecular-Weight — Heparin from start till hcg test
  Arms: Heparin, Low-Molecular-Weight group
Drug: no heparin
  Arms: Non Heparin, Low-Molecular-Weight group

SUMMARY:
The addition of heparin increases pregnancy outcome parameters in poor responders undergoing In Vitro Fertilisation (IVF)

ELIGIBILITY:
Inclusion Criteria:

* poor responders (age>40, abnormal ovarian test, </=4 oocytes in previous cycle with conventional stimulation)
* infertility, indication for IVF
* no contraindications for heparin

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
no of oocytes retrieved | egg recovery, 2 years
  >2 between groups

SECONDARY OUTCOMES:
clinical pregnancy rate | 2 years
  Presence of fetal heart at transvaginal ultrasound at 6+2 gestational weeks
live birth rate | 2 years
  >20 weeks of gestation
cancellation rate | before ET, 2 years
miscarriage rate | 2 years
  pregnancy loss <20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Department of Obstetrics & Gynecology, Athens, Chaidari, Greece